CLINICAL TRIAL: NCT02249637
Title: A Novel Technique of Circumcision Incision Orchidopexy for Palpable Low Inguinal Cryptorchidism: A Preliminary Report
Brief Title: A Novel Technique of Circumcision Incision Orchidopexy
Status: Completed | Type: Observational
Sponsor: St. Luke's Medical Center, Philippines (Other)
Collaborators: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Michael E. Chua, Urology Staff, St. Luke's Medical Center, Philippines
Other Study IDs: SLMC_2014(SLIU1)
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Cryptorchidism; Undescended Testis
MeSH Terms: conditions — Cryptorchidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Inguinal Orchidopexy: Patients with diagnosed palpable low inguinal cryptorchidism underwent inguinal approach as originally described by Schuller and Bevan.
- Novel Technique (Circumcision incision): Patients with diagnosed palpable low inguinal cryptorchidism underwent novel technique- circumcision incision orchidopexy.
  Interventions: Procedure: Novel technique Circumcision Incision Orchidopexy

INTERVENTIONS:
Procedure: Novel technique Circumcision Incision Orchidopexy — The novel technique starts with retraction of the prepucial skin off the glans penis and double incision circumcision done with mucosal sparing, then degloving of the penis on the side of the undescended testis. Dissection via Dartos' layer into the inguinal area until the palpable testicle was identified and extracted with mobilization of the spermatic cord. Hernia sac was then separated and suture ligated as high as the area of internal ring opening. Spematic cord lengthening was done until adequate length achieved for fixation into the inferior aspect of the scrotum. Then development of the Dartos' pouch via the circumcision site was done. A double or single suture testicular fixation using Vicryl 3-0 simple interrupted sutures on the everted Dartos' pouch inner surface was done. Subsequent placement of the testicle into the Dartos' pouch was done as the inner surface was inverted. The last step was the completion of the circumcision closure using Chromic 4-0 interrupted sutures.
  Other Names: Chua's Procedure
  Groups: Novel Technique (Circumcision incision)

SUMMARY:
Given that both circumcision and orchidopexy are commonly done in a single setting, the investigators adopted the technique of orchidopexy via circumcision incision, particularly for palpable low inguinal cryptorchidism. In this paper, the investigators aim to present a novel technique and discuss our preliminary outcome of such procedure compared to the traditional inguinal-scrotal double incision technique. Specifically, the investigators aimed to determine the differences in operative time, testicular size changes, peri-operative complications, pain score and parent's satisfaction of both novel technique and conventional orchidopexy.

DETAILED DESCRIPTION:
Cryptorchidism is the most common disorder of the male endocrine gland in children.. 1 According to the latest guideline by European Association of Urology in the Pediatric Urology for the treatment of cryptorchidism, both inguinal and scrotal approaches orchidopexy are accepted standard treatment options. 2 In the local setting, circumcision is another common surgical procedure among the children, particularly under the same instance of anesthesia for other procedure. Not only due to religious and sociocultural reasons, male circumcision has been recently considered having a protective effect against acquisition of various sexually transmitted infections (STIs). 3 This benefit is one of many that have led to many affirmative evidence-based policy statements by medical bodies in support of the procedure.

Given that both procedures are commonly done in a single setting, we adopted the technique of orchidopexy via circumcision incision, particularly for palpable low inguinal cryptorchidism. In this paper, we aim to present a novel technique and discuss our preliminary outcome of such procedure compared to the traditional inguinal-scrotal double incision technique. Specifically, we aimed to determine the differences in operative time, testicular size changes, peri-operative complications, pain score and parent's satisfaction of both novel technique and conventional orchidopexy.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with palpable cryptorchidism with pre-operative inguino-scrotal ultrasound to confirm the location of the testis on the low inguinal canal and its viability.

Exclusion Criteria:

* Excluded were non-palpable testis, with prior orchidopexy, circumcised, with other concomitant genital anomalies.

Ages: 3 Months to 10 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed with palpable cryptorchidism with pre-operative inguino-scrotal ultrasound to confirm the location of the testis on the low inguinal canal and its viability. Recruited from September 2013- September 2014
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Complication rate occurence related to the procedure | 3 months- 5 years
  Perioperative complications such as incidents of persistence of procesus vaginalis, testicular atrophy, hematoma, surgical site wound infection as well as the post-operative outcome such as testicular size changes

SECONDARY OUTCOMES:
Visual analogue scale (VAS) pain score post-operation | post-operative 24-48 hour
  Average pain score post operation as described by the patient using visual analogue scale
Parent's satisfaction score for the procedure post-operation | 1 week post operative follow up
  Parent's satisfaction score measured as 1-5 scale, with 1 being very unsatisfied, 2 being unsatisfied, 3 being neutral, 4 being satisfied, 5 being very satisfied
Operative time consumed by the procedure | Operative time
  Time from incision to incision closure end

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Urology, Quezon City, NCR, Philippines